CLINICAL TRIAL: NCT05104762
Title: IVIG Versus Plasmapheresis and Guillian Barrie Syndrome
Brief Title: IVIG Versus Plasmapheresis in the Treatment of Guillian Barrie Syndrome Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Guillian Barrie syndrome
Record Dates: First submitted 2021-10-21; First posted 2021-11-03 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Guillain-Barre Syndrome
Keywords: IVIG / plasmapheresis and Guillain-Barre Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: 2 groups of patients with Guillian Barrie syndrome were subjected to plasmapheresis or IVIG by percentage 2:1 respectively according to availability of IVIG
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind (participant and investigator, accessor) using closed envelope 2:1 was applied. 5 sessions of plasmapheresis: IVIG 0.4g IVIG/Kg /day for 5 consecutive days. The investigators didn't know what was the type of treatment that patients received and the patient didn't know that there is another line of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 plasmapheresis (Active Comparator): Arm 1 (plasmapheresis): This study will be conducted at Assiut University at Neurology and psychiatry department as Group 1 of patients presented with Guillian Barrie syndrome (54 patients) will be subjected to plasmapheresis after assessment of clinical state and scales including MRC, Erasmus Guillain-Barre respiratory insufficiency score and Overall neuropathy limitation scale and Neurophysiological studies. Each patient was evaluated at baseline and at Follow up assessment points (one month and 3 months, one year follow up)
  Interventions: Device: plasmapheresis device
- Arm 2: Intravenous injection of immunoglobulin (Active Comparator): This study will be conducted at Assiut University at Neurology and psychiatry department as Group 2 of patients presented with Guillian Barrie syndrome (27 patients) will be subjected to intravenous injection of immunoglobulin after assessment of clinical state and scales including MRC, Erasmus Guillain-Barre respiratory insufficiency score, and Overall neuropathy limitation scale and Neurophysiological studies. Each patient was evaluated at baseline and at Follow up assessment points (one month and 3 months, one year follow up).
  Interventions: Drug: Intravenous immunoglobulin

INTERVENTIONS:
Device: plasmapheresis device — Group 1: 54 patients of Guillian Barrie syndrome undergo plasma exchange (5 sessions)
  Other Names: plasma exchange device
  Arms: Arm 1 plasmapheresis
Drug: Intravenous immunoglobulin — group 2: 27 patients undergo intravenous injection of immunoglobulin for 5 consecutive days of IVIG 0.4gm/kg/day.
  Other Names: IVIG
  Arms: Arm 2: Intravenous injection of immunoglobulin

SUMMARY:
In this study, the investigators address the question: whether treatment with IVIG is superior to treatment using plasmapheresis for functional recovery of patients with GBS? Recovery was quantified using: The changes in the A-Clinical grading scale MRC ( medial research council sum score ) and B-overall neuropathy limitations scale as the primary outcome and the changes in Neurophysiological study 3 months after treatment as a secondary outcome.

This information will be used to evaluate which treatment is more beneficial to GBS patients.

DETAILED DESCRIPTION:
Guillain-Barré syndrome (GBS) is an inflammatory disease of the PNS and is the most common cause of acute flaccid paralysis, with an annual global incidence of approximately 1-2 per 100,000 person-years. Patients with GBS typically present with weakness and sensory signs in the legs that progress to the arms and cranial muscles, although the clinical presentation of the disease is heterogeneous and several distinct clinical variants exist. Diagnosis of GBS is based on the patient's history and neurological, electrophysiological, and cerebrospinal fluid (CSF) examinations. Electrophysiological studies: provide evidence of peripheral nervous system (PNS) dysfunction and can distinguish between the subtypes of GBS: acute inflammatory demyelinating polyradiculoneuropathy (AIDP), acute motor axonal neuropathy (AMAN), and acute motor-sensory axonal neuropathy (AMSAN). Disease progression can be rapid, and most patients with GBS reach their maximum disability within 2 weeks. About 20% of patients with GBS develop respiratory failure and require mechanical ventilation. Cardiac arrhythmias and blood pressure instability can occur owing to the involvement of the autonomic nervous system. Immunomodulatory therapy should be started if patients are unable to walk independently for 10 m. Evidence on treatment efficacy in patients who can still walk independently is limited, but treatment should be considered, especially if these patients display rapidly progressive weakness or other severe symptoms such as autonomic dysfunction, bulbar failure, or respiratory insufficiency. Clinical trials have demonstrated a treatment effect for intravenous immunoglobulin (IVIg) when started within 2 weeks of the onset of weakness and for plasma exchange when started within 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years old,
* Onset: Recent onset of GBS through the first 2 weeks.
* Gender: Male or Female Inclusion Criteria.

Exclusion Criteria:

* patients with metabolic disorders, or malignancy,
* other causes of peripheral neuropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Clinical grading scale MRC ( medial research council sum score ) | the points change from baseline scale and after 3 months follow up
  Clinical grading scale MRC ( medial research council sum score ) from zero ( no power ) up to 60 full power (points): sum score of muscle power in both upper limbs and lower limbs in points .
Overall neuropathy limitations scale (ONLS) . | the changes in points from baseline assessment score to 3 months follow up assessment score.
  it is modified disability sum score: sum of arm grade and leg grade limitation score; arm grade from zero point ( less limitation ) to 5 points ( most limitation ) and leg grade from zero point ( less limitation) to 7 points (more limitation)
ERASMUS GBS respiratory insufficiency score EGRIS | the change in points from baseline assessment score to 3 months follow up assessment score.
  Predict the probability of respiratory insufficiency within the first week of admission, in individual patients with Guillain-Barre. syndrome from zero to 7 points score : 0 point ( no affection ) , 7 point ( severe affection )

SECONDARY OUTCOMES:
Neurophysiological study: Distal latency in mill second, Nerve conduction velocities in Meter/second, and F-wave latency mill second | the change in points from baseline assessment score to 3 months follow up assessment score.
  Neurophysiological study neurophysiological study pre- and after 3 months change of degree of affection and improvement in latency in nerve conduction m/ sec. amplitude m/v , velocity of nerve /s conduction and F-wave of both upper limbs and lower limbs

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Dornonville de la Cour C, Jakobsen J. Residual neuropathy in long-term population-based follow-up of Guillain-Barre syndrome. Neurology. 2005 Jan 25;64(2):246-53. doi: 10.1212/01.WNL.0000149521.65474.83. PMID 15668421
- [Background] van Koningsveld R, Steyerberg EW, Hughes RA, Swan AV, van Doorn PA, Jacobs BC. A clinical prognostic scoring system for Guillain-Barre syndrome. Lancet Neurol. 2007 Jul;6(7):589-94. doi: 10.1016/S1474-4422(07)70130-8. PMID 17537676
- [Background] Fokke C, van den Berg B, Drenthen J, Walgaard C, van Doorn PA, Jacobs BC. Diagnosis of Guillain-Barre syndrome and validation of Brighton criteria. Brain. 2014 Jan;137(Pt 1):33-43. doi: 10.1093/brain/awt285. Epub 2013 Oct 26. PMID 24163275
- [Background] Walgaard C, Lingsma HF, Ruts L, van Doorn PA, Steyerberg EW, Jacobs BC. Early recognition of poor prognosis in Guillain-Barre syndrome. Neurology. 2011 Mar 15;76(11):968-75. doi: 10.1212/WNL.0b013e3182104407. PMID 21403108
- [Background] Raphael JC, Chevret S, Hughes RA, Annane D. Plasma exchange for Guillain-Barre syndrome. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD001798. doi: 10.1002/14651858.CD001798.pub2. PMID 22786475
- [Background] van Doorn PA, Ruts L, Jacobs BC. Clinical features, pathogenesis, and treatment of Guillain-Barre syndrome. Lancet Neurol. 2008 Oct;7(10):939-50. doi: 10.1016/S1474-4422(08)70215-1. PMID 18848313
- [Background] van Doorn PA. Diagnosis, treatment and prognosis of Guillain-Barre syndrome (GBS). Presse Med. 2013 Jun;42(6 Pt 2):e193-201. doi: 10.1016/j.lpm.2013.02.328. Epub 2013 Apr 28. PMID 23628447
- [Background] van Nes SI, Vanhoutte EK, van Doorn PA, Hermans M, Bakkers M, Kuitwaard K, Faber CG, Merkies IS. Rasch-built Overall Disability Scale (R-ODS) for immune-mediated peripheral neuropathies. Neurology. 2011 Jan 25;76(4):337-45. doi: 10.1212/WNL.0b013e318208824b. PMID 21263135
- [Background] Mori M, Kuwabara S, Fukutake T, Hattori T. Intravenous immunoglobulin therapy for Miller Fisher syndrome. Neurology. 2007 Apr 3;68(14):1144-6. doi: 10.1212/01.wnl.0000258673.31824.61. PMID 17404197
- [Background] Kalita J, Misra UK, Goyal G, Das M. Guillain-Barre syndrome: subtypes and predictors of outcome from India. J Peripher Nerv Syst. 2014 Mar;19(1):36-43. doi: 10.1111/jns5.12050. PMID 24456386